CLINICAL TRIAL: NCT02303236
Title: Biological Markers Predicting Exercise Capacity in Heart Failure Patients Supported With a Continuous-flow Left Ventricular Assist Device.
Brief Title: Biological Markers Predicting Exercise Capacity in CF-LVAD Patients.
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Finn Gustafsson, MD, Ph.D, Rigshospitalet, Denmark
Other Study IDs: H-1-2012-092-B
Record Dates: First submitted 2014-11-20; First posted 2014-11-27 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Heart Failure
Keywords: Exercise
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples in biological bank.
Oversight: Data Monitoring Committee: No

SUMMARY:
Establishing the association between biological markers and exercise capacity in continuous-flow left ventricular assist device patients.

DETAILED DESCRIPTION:
The aim of this study is to investigate if specific biological markers can predict exercise capacity in advanced heart failure patients supported with continuous-flow left ventricular assist device patients.

ELIGIBILITY:
Inclusion Criteria:

* Stable CF-LVAD patients.

Exclusion Criteria:

* Unstable CF-LVAD patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable CF-LVAD patients.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12-24 (Actual)

PRIMARY OUTCOMES:
Biological markers | Blood sampling on study day and samples are subsequently stored frozen.
  Analysis of blood will be carried out on all samples simultaneously, expected markers are pro-BNP, MRproANP, copeptin, Gal-3 and proADM.

SECONDARY OUTCOMES:
Exercise capacity | Examination on study day. Patients will only be followed on the day of the study. Exercise testing is performed as the last intervention on the study day.
  Exercise capacity will be estimated by peak VO2 measurements on a upright ergometer bike with breath-by-breath gas analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gustafsson, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- University Hospital Rigshospitalet., Copenhagen, Kbh Oe, Denmark